CLINICAL TRIAL: NCT01247805
Title: A Pivotal Randomised, Open-Label 3-Way Crossover Study To Demonstrate Bioequivalence Of The Sildenafil Citrate Powder For Oral Suspension (10 Mg/Ml) And The Sildenafil Citrate 10 Mg Immediate Release (IR) Tablet Relative To The Revatio 20 Mg IR Tablet In Healthy Volunteers Under Fasting Conditions
Brief Title: A Pivotal Bioequivalence Study Between The Sildenafil Powder For Oral Suspension (10 Mg/Ml) And The Sildenafil 10 Mg Immediate Release (IR) Tablet Relative To The Revatio 20 Mg IR Tablet In Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A1481293; EudraCT 2010-023521-38
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertention
Keywords: Bioequivalence; Powder for oral suspention
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Revatio: 1 x 20 mg IR oral tablet.
  Interventions: Drug: sildenafil citrate
- Treatment B (Experimental): 2 x 10 mg sildenafil citrate IR oral tablet.
  Interventions: Drug: Sildenafil citrate
- Treatment C (Experimental): 2 mL of the 10 mg/mL sildenafil citrate POS (20 mg dose).
  Interventions: Drug: sildenafil citrate

INTERVENTIONS:
Drug: sildenafil citrate — Single oral dose of 1 x 20 mg IR oral tablet.
  Other Names: Revatio
  Arms: Treatment A
Drug: Sildenafil citrate — single oral dose of 2 x 10 mg sildenafil citrate IR oral tablet.
  Other Names: Revatio
  Arms: Treatment B
Drug: sildenafil citrate — single oral dose of 2 mL of the 10 mg/mL sildenafil citrate POS (20 mg dose).
  Other Names: Revatio
  Arms: Treatment C

SUMMARY:
The hypothesis for the trial is that the Sildenafil Citrate Powder for Oral Suspension (10 Mg/ml) bioequivalent to the Revatio 20 Mg IR tablet in Healthy Volunteers and the Sildenafil Citrate 10 Mg immediate release (IR) tablet is bioequivalent to the Revatio 20 Mg IR tablet in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

1) Healthy male/female subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests.

2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

3. An informed consent document signed and dated by the subject or a legally acceptable representative.

4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, ocular or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing) disease or clinical findings at Screening.
2. History of febrile illness within 5 days prior to the first dose.
3. A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC0-T) of sildenafil plasma concentrations from time zero to the time T of last measurable concentration. | Pre-dose, 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 14 hours post dose
Maximum sildenafil plasma concentration (Cmax) | Pre-dose, 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 14 hours post dose

SECONDARY OUTCOMES:
AUCinf, AUC of sildenafil from time zero to time infinity. AUCinf = AUC0-T+AUCextrapolated | Pre-dose, 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 14 hours post dose
AUC%extrapolated of sildenafil. | Pre-dose, 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 14 hours post dose
Tmax - time at which maximum sildenafil plasma concentration occurs | Pre-dose, 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 14 hours post dose
Adverse events | From FSFV to LSLV, up to 5 weeks
terminal half-life of sildenafil. | Pre-dose, 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 14 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481293&StudyName=A%20Pivotal%20Bioequivalence%20Study%20Between%20The%20Sildenafil%20Powder%20For%20Oral%20Suspension%20%2810%20Mg/Ml%29%20And%20The%20Sildenafil%2010%20Mg%20Immediate%20Relea